CLINICAL TRIAL: NCT01829958
Title: Comprehensive Geriatric Assessment to Predict Toxic Events in Older Patients With Non-Hodgkin Lymphoma With Imbedded Pilot Study of Pre-Phase Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-028
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma (NHL); Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Geriatric; Toxicity; rituximab; prednisone; Comprehensive Geriatric Assessment (CGA); 13-028
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Prednisone; Geriatric Assessment

ARMS (2):
- Pre-Phase Arm (Experimental): They will be treated with a single dose of rituximab 375mg/m2, once, by intravenous infusion 3-10 days prior to initiation of planned R-CHOP-like chemoimmunotherapy, and prednisone 50mg to 100 mg (preferred dose is 100mg) PO daily for 5-7 days (preferred duration is 7 days) of the 14 days prior to initiation of planned R-CHOP, R-EPOCH or R-CEPP chemoimmunotherapy. Pre-phase therapy may be given in either the inpatient or outpatient setting. After completion of a single course of pre-phase rituximab and prednisone as described above, further treatment will be according to the choice of the attending physician, in accordance with appropriate medical practice. It is expected, based on the inclusion criteria, that patients enrolled on the pre-phase arm will most often receive initial therapy consisting of R-CHOP, R-EPOCH or RCEPP chemoimmunotherapy for ≥ 2 cycles, but alternative therapies as deemed appropriate by the treating physician will not be considered violations of this protocol.
  Interventions: Drug: rituximab; Drug: prednisone; Behavioral: Geriatric Assessment
- Geriatric Assessment (GA) only arm (Experimental): Patients enrolled on the GA only arm of the study will be treated according to the choice of the attending physician. This arm of the study is non-therapeutic.
  Interventions: Behavioral: Geriatric Assessment

INTERVENTIONS:
Drug: rituximab
  Arms: Pre-Phase Arm
Drug: prednisone
  Arms: Pre-Phase Arm
Behavioral: Geriatric Assessment

SUMMARY:
This study will evaluate the ability of a largely self-administered geriatric assessment (GA) to predict toxicity in non-Hodgkin Lymphoma (NHL) patients ≥60 years old receiving chemotherapy or chemoimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria will be eligible for enrollment in the study (unless excluded):

* ≥60 years old
* Pathologically confirmed NHL.
* Must meet criteria for initiation of treatment; consisting of:
* Aggressive histology, or
* Indolent histology with one of the following markers of large tumor burden (67):
* Any nodal or extranodal tumor mass ≥7cm in greatest dimension
* ≥3 nodal masses that are each ≥3 cm in greatest dimension
* Systemic symptoms
* Cytopenias (leukocytes <1 × 109/L and/or platelets ,100 × 109/L)
* Substantial splenomegaly
* Serous effusion (plural effusion or peritoneal ascites)
* Orbital or epidural involvement
* Ureteral compression
* Leukemic phase (malignant cells ≥5 x 109/L)
* Must be starting a new chemotherapy regimen (patients whose treatment regimen includes an immunomodulatory agent such as lenalidomide or small molecule targeted agents such as Ibrutinib or Idelelasib will be included in the study; patients being treated with a single agent monoclonal antibody will not be included).
* Fluent in English (because not all components of the GA have been validated in other languages)
* Able to provide informed consent

In addition to the above, subjects meeting the following criteria will be enrolled in the pre-phase arm of the study, until the accrual target for that arm is reached:

* Age ≥ 70 years OR KPS ≤ 70
* Pathologically confirmed diagnosis of DLBCL, with or without simultaneous or antecedent indolent lymphoma.
* Previously untreated for DLBCL
* Intended initial treatment to include ≥2 cycles of R-CHOP, R-EPOCH or R-CEPP using standard doses and schedule.(68, 69) R-CHOP chemoimmunotherapy may be given every 14 days or every 21 days. (4, 70)

Exclusion Criteria:

Subjects meeting the following criteria will be excluded from enrollment in the study:

* Enrollment in a Phase I trial
* Previously enrollment in this study
* Patients scoring ≥ 11 on the BOMC (implying cognitive impairment) will be excluded since their ability to reliably complete the questionnaire will be in doubt Subjects meeting the following criteria will be excluded from enrollment in the pre-phase arm of the study, but may be included in the GA only arm.
* Contraindication to use of rituximab or prednisone including:
* Uncontrolled diabetes mellitus
* Systemic fungal infection
* Evidence of active hepatitis B infection (i.e. patients testing positive hepatitis B surface antigen or viral DNA by PCR analysis) will be excluded. Patients with evidence of past infection without active viremia (i.e. positive hepatitis B core antibody, negative hepatitis B surface antigen and negative hepatitis B DNA PCR) will be treated with entecavir as per institutional guidelines and may be included in the study.
* History of any serious adverse reaction to either a corticosteroid or rituximab not including rituximab infusion reactions ≤ Grade 3.
* Patients enrolled on another clinical trial which prohibits the use of pre-phase therapy or any of its components.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Toxicity Assessment | 3 years
  Hospitalization during or within 30 days following chemotherapy Dose delay or reduction to a dose intensity ≤80% of the planned dose intensity. Dose reductions occurring prior to cycle 1 of chemotherapy will be counted as events. Discontinuation of chemotherapy due to toxicity Grade 3 or higher non-hematologic toxicity Grade 4 or higher hematologic toxicity. Using the NCI CTCAE v4.0 toxicity grading

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hamlin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/